CLINICAL TRIAL: NCT00880997
Title: Doxazosin, An Alpha-1 Adrenergic Antagonist, for Cocaine Dependence: Pilot Study
Brief Title: The Efficacy of Doxazosin for Cocaine Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Thomas R. Kosten, MD, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-18197-4; P50DA018197-04 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Cocaine Dependence
Keywords: Cocaine Dependence; Substance Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Doxazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxazosin (Experimental): Medication induction occurred at a rate of 2mg/week until 8mg/day target dose was achieved as follows:
  1. Dox-Fast Group: Defined as participants reaching the target dose after a 4-week titration period. Participants were stabilized on doxazosin or placebo over weeks 4-13 (for Dox-Fast group)
  2. Dox-Slow Group: Defined as participants reaching the target dose after an 8-week titration period. Participants were stabilized on doxazosin or placebo over weeks 8-13 (for Dox-Slow group)
  Both groups were tapered off doxazosin or placebo over study weeks 14-17.
  Interventions: Drug: Doxazosin
- placebo (Placebo Comparator): A sugar pill to mimic the experiment drug, doxazosin, will be administered in the same manner as the experimental drug through the study duration.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Doxazosin — Medication induction occurred at a rate of 2mg/week until 8mg/day target dose was achieved as follows:
  1. Dox-Fast Group: Defined as participants reaching the target dose after a 4-week titration period. Participants were stabilized on doxazosin or placebo over weeks 4-13 (for Dox-Fast group)
  2. Dox-Slow Group: Defined as participants reaching the target dose after an 8-week titration period. Participants were stabilized on doxazosin or placebo over weeks 8-13 (for Dox-Slow group)
  Both doxazosin groups will be tapered off doxazosin or placebo over study weeks 14-17.
  Other Names: Cardura (Doxazosin Mesylate)
  Arms: Doxazosin
Other: Placebo — Participants will be administered a sugar pill to mimic the doxazosin active medication with administration being the same as the active medication.
  Other Names: sugarpills ( Capsules)
  Arms: placebo

SUMMARY:
Doxazosin, an alpha 1-adrenergic receptor, may play an important role in cocaine addiction in humans. This study will evaluate the effectiveness of doxazosin in preventing drug relapse among cocaine dependent participants.

DETAILED DESCRIPTION:
The NE system, especially the alpha 1-adrenergic receptor, may play an important role in cocaine addiction in humans. The results of this study will provide medical safety data on the duration of the induction schedule that will be optimal for attaining our target dose of 8 mg doxazosin daily and will guide future pharmacotherapy trials using Doxazosin or related alpha 1 receptor antagonists for cocaine addiction.

This 17-week double-blind, placebo controlled clinical trial includes a 13 week medication trial (weeks 1-13) and up to 4 week washout period(weeks 14-17). Qualifying subjects will be randomized to receive Doxazosin 8 mg/day, or placebo during the study participation.

Medication induction will occur at a rate of 2mg/week until 8mg/day target dose is achieved as follows:

1. Dox-Fast Group: Defined as participants reaching the target dose after a 4-week titration period. Participants will be stabilized on doxazosin or placebo over weeks 4-13 (for Dox-Fast group)
2. Dox-Slow Group: Defined as participants reaching the target dose after an 8-week titration period. Participants will be stabilized on doxazosin or placebo over weeks 8-13 (for Dox-Slow group)

Both groups will be tapered off doxazosin or placebo over study weeks 14-17.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV diagnosis criteria for cocaine dependence, as determined by self-reported use of cocaine at least once weekly for at least 1 month prior to study entry; a positive urine test for cocaine; and a score greater than 3 on the Severity of Dependence Scale
* If female, willing to use contraception throughout the study

Exclusion Criteria:

* Meets DSM-IV diagnosis criteria for dependence on any drugs other than cocaine, or tobacco
* Current major psychiatric illness, including schizophrenia, bipolar disorder, or other psychotic disorder
* Current suicidal or homicidal ideation
* Current use of a prescribed psychotropic medication that cannot be discontinued
* History of or current major medical illness, including major heart, kidney, endocrine, or liver disorder; abnormal liver function (SGOT or SGPT levels three times greater than normal); or high blood pressure or low blood pressure
* High risk factor for heart disease, seizure disorders, or any illness for which disulfiram or methadone treatment would be inadvisable
* Currently taking metronidazole or clotrimazole
* Pregnant or breastfeeding

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Kosten, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine - Michael E. DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-five subjects were randomized into the study, with 30 subjects returning and receiving at least one dose of medication.
Groups:
- Doxazosin Fast: Participantsreaching the target dose after a 4-week titration period
- Doxazosin Slow: Participants reaching the target dose after an 8-week titration period
- Placebo: Matching placebo
Period: Overall Study
Arm/Group | Doxazosin Fast | Doxazosin Slow | Placebo
Started | 9 | 8 | 13
Completed | 6 | 6 | 5
Not Completed | 3 | 2 | 8

BASELINE CHARACTERISTICS:
Population: Cocaine dependent individuals = 17; Placebo = 13; 5 lost to followup. During analysis, an additional 2 individuals were dropped due from analyses due to invalidated data.
Groups:
- Doxazosin Slow Titration: Medication induction occurred at a rate of 2mg/week until 8mg/day target dose was achieved as follows:
  Dox-Slow Group: Participants reaching the target dose after an 8-week titration period. Participants were stabilized on doxazosin over weeks 8-13.
  Participants were tapered off doxazosin or placebo over study weeks 14-17.
- Doxazosin Fast Titration: Medication induction occurred at a rate of 2mg/week until 8mg/day target dose was achieved as follows:
  Dox-Fast Group: Participants reaching the target dose after a 4-week titration period. Participants were stabilized on doxazosin over weeks 4-13.
  Participants were tapered off doxazosin or placebo over study weeks 14-17.
- Placebo: Participants received matched placebo during weeks 1-13.
  Participants were tapered off placebo over study weeks 14-17.
- Total: Total of all reporting groups
Arm/Group | Doxazosin Slow Titration | Doxazosin Fast Titration | Placebo | Total
Number analyzed (Participants) | 8 | 9 | 13 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 13 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (7.4) | 47.4 (11.0) | 48.2 (8.6) | 48 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 4
  Male | 8 | 7 | 11 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 3 | 10 | 20
  White | 1 | 6 | 3 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 13 | 30
Employment [Count of Participants; unit: Participants] — Employed over the past 3 years
  Participants | 6 | 7 | 9 | 22
Alcohol use - past 30 days [Mean (Standard Deviation); unit: days] | 6.63 (3.77) | 10.11 (9.55) | 7.85 (9.89) | 8.5 (8)
Cocaine use - past 30 days [Mean (Standard Deviation); unit: days] | 18.13 (8.90) | 7.89 (6.92) | 14.85 (10.25) | 15 (8.27)

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Negative Urines
Description: cocaine urine toxicology samples were obtained thrice weekly and tested for the presence of the cocaine metabolite, benzoylecgonine
Time Frame: throughout the study - up to 17 weeks
Measure: Number; unit: percentage of cocaine-negative urines
Groups:
- DOX-slow Group: Participants reaching the target dose after an 8-week titration period are labeled as the DOX slow group. Participants were stabilized on doxazosin over weeks 8-13 and then tapered off doxazosin over study weeks 14-17.
- DOX-fast Group: Participants reaching the target dose after a 4-week period are labeled as the DOX-fast group. Participants were stabilized on doxazosin over weeks 4-13 and then tapered off doxazosin over study weeks 14-17.
- Placebo: Participants took placebo during weeks 1-17.
Arm/Group | DOX-slow Group | DOX-fast Group | Placebo
Number analyzed (Participants) | 8 | 9 | 13
percentage of cocaine-negative urines | 10 | 35 | 14

2. Secondary Outcome: Weeks of Abstinence
Description: Percentage of participants achieving 2 or more consecutive weeks of abstinence
Time Frame: throughout the study - up to 17 weeks
Measure: Number; unit: percentage of participants
Arm/Group | DOX-slow Group | DOX-fast Group | Placebo
Number analyzed (Participants) | 8 | 9 | 13
percentage of participants | 0 | 44 | 7

3. Secondary Outcome: # of Participants That Completed the Study
Description: Retention
Time Frame: throughout the study - up to 17 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | DOX-slow Group | DOX-fast Group | Placebo
Number analyzed (Participants) | 8 | 9 | 13
Participants | 6 | 6 | 5

4. Secondary Outcome: Adverse Events
Time Frame: throughout study - upto 17 weeks
Measure: Number; unit: events
Arm/Group | DOX-slow Group | DOX-fast Group | Placebo
Number analyzed (Participants) | 8 | 9 | 13
events | 26 | 9 | 23

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the entire study duration for all patients, up to 17 weeks.
Groups:
- Dox-Slow Group: Defined as participants reaching the target dose after an 8-week titration period. Participants were stabilized on doxazosin or placebo over weeks 8-13 (for Dox-Slow group)
- Dox-Fast Group:: Defined as participants reaching the target dose after a 4-week titration period. Participants were stabilized on doxazosin or placebo over weeks 4-13 (for Dox-Fast group)
- Placebo: A sugar pill to mimic the experiment drug, doxazosin, will be administered in the same manner as the experimental drug through the study duration.
  Placebo: Placebo daily dosing
Arm/Group | Dox-Slow Group | Dox-Fast Group: | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/13
Other Adverse Events (participants affected / at risk) | 2/8 | 3/9 | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dox-Slow Group (N=8) | Dox-Fast Group: (N=9) | Placebo (N=13)
Headaches (Nervous system disorders) | 2 | 1 | 3
Dizinness (Cardiac disorders) | 0 | 2 | 0
Toothache (General disorders) | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
Initially the study randomized subjects into 2 conditions (placebo/DOX). After the observation that rapid titration was safe, a DOX-fast group was created. This did not allow for early participants to be randomized to the rapid titration condition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No